CLINICAL TRIAL: NCT07329335
Title: Comparison of High-Intensity Interval Training and Medium-Intensity Interval Training on Cardiopulmonary Fitness, Strength and Agility in Athletes
Brief Title: Comparison of High-Intensity Interval Training and Medium-Intensity Interval Training in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0479
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Athletes
Keywords: High Intensity Training , Medium Intensity Training , Athletes

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (High Intensity interval Training) (Experimental): Group A (High Intensity interval Training) Group A will engage in a structured High-Intensity Interval Training (HIIT) program over a 6-week period, with sessions to enhance cardiopulmonary fitness, strength, and agility.
  Interventions: Other: High Intensity Training (Group A)
- Group B (Moderate Intensity Interval Training): (Experimental): Group B (Moderate Intensity Interval Training):
  Group B will participate in a structured Medium-Intensity Interval Training (MIIT) program over a 6-week period, with sessions aimed at gradually improving endurance, strength, and coordination.
  Interventions: Other: Medium Intensity Training (Group B)

INTERVENTIONS:
Other: High Intensity Training (Group A) — Each 45-minute session will begin with a 5-minute warm-up consisting of dynamic stretches targeting major muscle groups. The main workout will include high-intensity cardio intervals, strength exercises, and agility drills, such as sprints, jump squats, and ladder drills, performed in short bursts with brief rest periods. The session will end with a cool-down phase of static stretching to support recovery and flexibility.
  Arms: Group A (High Intensity interval Training)
Other: Medium Intensity Training (Group B) — Each 45-minute session will start with a 5-minute warm-up of dynamic stretches. The main workout will start with moderate-paced cardio intervals, strength exercises, and agility drills, such as jogging, bodyweight squats, and cone drills, allowing for steady effort with manageable rest intervals. The session will end with a cool-down phase of static stretching to promote muscle recovery and flexibility.
  Arms: Group B (Moderate Intensity Interval Training):

SUMMARY:
High-Intensity Interval Training (HIIT) and Medium-Intensity Interval Training (MIIT) are popular training methods known for enhancing athletic performance. HIIT is characterized by short bursts of high-intensity exercise followed by brief recovery periods. This training approach typically involves exercising at 80-95% of maximum heart rate for intervals ranging from 20 seconds to a few minutes, followed by rest or lower-intensity activity. Moderate-Interval Training (MIIT), on the other hand, involves moderate-intensity exercise performed at 60-75% of maximum heart rate. The primary objective is to determine how HIIT and MIIT differ in improving CPF, strength, and agility among athletes. A randomized clinical trial will be conducted with a sample size of 80 athletes, divided into two groups. Participants will undergo 45-minute training sessions three times a week for six weeks, followed by pre- and post-intervention assessments using Cooper's 12-Minute Run/Walk Test, T-Test for agility, and Active Force 2 muscle tester for strength. Statistical analyses will be conducted to compare pre- and post-intervention results between the two groups, determining the significance of differences in CRF fitness, strength and agility outcomes.

DETAILED DESCRIPTION:
Study Design: Randomized Clinical Trial Sample size 72 (36 in each group)

Inclusion Criteria:

* Age 20-30 years
* Both male and female
* Athletes with BMI 18.5kg/m2 -24.9kg/m2 (14)
* Minimum 3 years of regular training in sports (20)

Exclusion Criteria:

* History of Any fracture or trauma (21)
* Having any neurological disease (21)
* Any chronic musculoskeletal disorder (21)
* Any systemic illnesses (21)
* Exclude athletes with known sleep disorders(e.g, insomnia ,sleep and apnoea )
* Athletes having consumption of pharmaceutical drugs e.g Beta blockers, benzodiazepines will be excluded

Data Collection Tools

1. Cooper's 12 minutes run/walk test (For Cardio respiratory Fitness)ICC 9.90
2. T test Agility (For Agility)ICC 0.75
3. Active Force 2 (For Strength) ICC 0.86-0.95

ELIGIBILITY:
Inclusion Criteria:

* Age 20-30 years
* Both male and female
* Athletes with BMI 18.5kg/m2 -24.9kg/m2
* Minimum 3 years of regular training in sports

Exclusion Criteria:

* History of Any fracture or trauma
* Having any neurological disease
* Any chronic musculoskeletal disorder
* Any systemic illnesses
* Exclude athletes with known sleep disorders(e.g, insomnia ,sleep and apnoea )
* Athletes having consumption of pharmaceutical drugs e.g Beta blockers, benzodiazepines will be excluded

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Cooper's 12 minutes run/walk test | 6 weeks
  Cooper's 12 minutes run/walk test (For Cardio respiratory Fitness) The Cooper 12 minute run is a popular maximal running test of aerobic fitness, in which participants try and cover as much distance as they can in 12 minutes. equipment required: flat oval or running track, marker cones, recording sheets, stop watch with a validity of 0.90.
T test Agility (For Agility) | 6 weeks
  T test Agility (For Agility) The T-test for agility is a reliable and valid measure to assess an individual's quickness and directional change ability. To ensure reliability, the test should be administered multiple times (test-retest reliability) and checked for consistent scoring between trials, ideally resulting in an Intraclass Correlation Coefficient (ICC) above 0.75, which indicates good reliability. Additionally, inter-rater and intra-rater reliability should be examined if multiple evaluators are involved.
Active Force 2 (For Strength) | 6 week
  Active Force 2 (For Strength) The Active Force 2 has demonstrated strong validity and reliability in muscle strength assessments. Its concurrent validity is high, with correlation coefficients ranging from 0.86 to 0.95 compared to established dynamometers, and construct validity values above 0.85 align with theoretical expectations for muscle strength measurements. Test-retest reliability values are robust, with intra class correlation coefficients (ICCs) between 0.92 and 0.98, indicating consistency across repeated measures. Additionally, intra-rater reliability ICCs range from 0.90 to 0.96, and inter-rater reliability ICCs from 0.88 to 0.95, reflecting consistent results when measurements are taken by the same or different testers.

CONTACTS AND LOCATIONS:
Overall Officials: Surakhsha Shaker, DPT, Principal Investigator — Riphah International University
Locations (1):
- Hafeez qadeer Cricket Academy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arboleda-Serna VH, Feito Y, Patino-Villada FA, Vargas-Romero AV, Arango-Velez EF. Effects of high-intensity interval training compared to moderate-intensity continuous training on maximal oxygen consumption and blood pressure in healthy men: A randomized controlled trial. Biomedica. 2019 Sep 1;39(3):524-536. doi: 10.7705/biomedica.4451. PMID 31584766
- [Background] Wen D, Utesch T, Wu J, Robertson S, Liu J, Hu G, Chen H. Effects of different protocols of high intensity interval training for VO2max improvements in adults: A meta-analysis of randomised controlled trials. J Sci Med Sport. 2019 Aug;22(8):941-947. doi: 10.1016/j.jsams.2019.01.013. Epub 2019 Jan 29. PMID 30733142
- [Background] Pereira PE, Esteves G, Carvas N, Azevedo PH. Effects of high-intensity interval and moderate-intensity continuous training on the anaerobic threshold of highly trained athletes in endurance sports: a systematic review with meta-analysis. J Sports Med Phys Fitness. 2024 Sep;64(9):898-907. doi: 10.23736/S0022-4707.24.15855-0. Epub 2024 Jun 6. PMID 38842374
- [Background] Guo Z, Li M, Cai J, Gong W, Liu Y, Liu Z. Effect of High-Intensity Interval Training vs. Moderate-Intensity Continuous Training on Fat Loss and Cardiorespiratory Fitness in the Young and Middle-Aged a Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2023 Mar 8;20(6):4741. doi: 10.3390/ijerph20064741. PMID 36981649
- [Background] Wang Z, Wang J. The effects of high-intensity interval training versus moderate-intensity continuous training on athletes' aerobic endurance performance parameters. Eur J Appl Physiol. 2024 Aug;124(8):2235-2249. doi: 10.1007/s00421-024-05532-0. Epub 2024 Jun 21. PMID 38904772
- [Background] Ballesta-Garcia I, Martinez-Gonzalez-Moro I, Rubio-Arias JA, Carrasco-Poyatos M. High-Intensity Interval Circuit Training Versus Moderate-Intensity Continuous Training on Functional Ability and Body Mass Index in Middle-Aged and Older Women: A Randomized Controlled Trial. Int J Environ Res Public Health. 2019 Oct 30;16(21):4205. doi: 10.3390/ijerph16214205. PMID 31671584